CLINICAL TRIAL: NCT02276937
Title: DVC1-0101 for Intermittent Claudication Secondary to Peripheral Artery Disease: a Randomized Phase IIb Trial
Brief Title: Randomized Phase IIb Trial of DVC1-0101
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kyushu University (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government); Japan Agency for Medical Research and Development (Other Government)
Responsible Party: Principal Investigator, Yoshikazu Yonemitsu, Professor, Kyushu University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTR-001; UMIN000014926 (Registry Identifier: UMIN CTR)
Record Dates: First submitted 2014-10-22; First posted 2014-10-28 (Estimated); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Intermittent Claudication; Peripheral Arterial Disease
Keywords: Recombinant Sendai virus; fibroblast growth factor-2; treadmill
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (0 ciu/limb) (Placebo Comparator): Placebo control
  Interventions: Drug: DVC1-0101
- DVC1-0101 low dose (1x10^9 ciu/limb) (Active Comparator): Low dose cohort
  Interventions: Drug: DVC1-0101
- DVC1-0101 high dose (5x10^9 ciu/limb) (Active Comparator): High dose cohort
  Interventions: Drug: DVC1-0101

INTERVENTIONS:
Drug: DVC1-0101 — The investigational product will be drawn into a disposable 1 mL syringe using a 23G needle. A total of 0.5 mL of investigational product will be injected intramuscularly into each administration site. After administration, the administration sites will be wrapped with dressings.
  Other Names: rSeV/dF expressing human FGF-2 gene

SUMMARY:
DVC1-0101 is a gene therapy medicine to treat peripheral arterial disease (PAD) based on recombinant F-gene-deleted, non-transmissible Sendai virus (rSeV/dF) expressing human fibroblast growth factor-2 (FGF-2) gene.

The primary objective of the current Phase IIb study is to investigate the clinical efficacy of DVC1-0101 (1x10^9 ciu/leg, 5x10^9 ciu/leg) in patients with IC.

DETAILED DESCRIPTION:
DVC1-0101 is a gene therapy medicine to treat peripheral arterial disease (PAD) based on recombinant F-gene-deleted, non-transmissible Sendai virus (rSeV/dF) expressing human fibroblast growth factor-2 (FGF-2) gene. The previous Phase I/IIa study demonstrated no serious adverse event related to the administration, and suggested possible improvement of local blood flow and walking performance of PAD patients.

The primary objective of the current Phase IIb study is to investigate the clinical efficacy of DVC1-0101 (1x10^9 ciu/leg, 5x10^9 ciu/leg) in patients with IC. We also aim to examine the dose-response relationship using the rate of improvement in walking function as an indicator.

ELIGIBILITY:
Inclusion Criteria:

1) Meet criteria (1) to (5) below and are confirmed as such by at least 1 specialist qualified by the Japanese Society for Cardiovascular Surgery and at least 1 physician with deep experience Cardiovascular Intervention.

1. arteriosclerosis obliterans with stable symptoms, have intermittent claudication (ACD < 260 m) and are able to walk on a treadmill
2. resting ankle-brachial pressure index < 0.9
3. refuse revascularization, risk of revascularization may be greater than the benefit, or develop obliteration after revascularization
4. angiographic findings show patency from the abdominal aorta through to the proximal side of the external iliac artery
5. angiographic findings meet the above criterion (4), and have stenosis or obliteration under the femoropopliteal region with morphology defined as type C or D based on TASCII

2) Administering cilostazol for at least 1 month and still meet criterion 1).

3) Aged 30 and over.

4) Either sex, either inpatients or outpatients.

5) Able to give written consent for themselves.

Exclusion Criteria:

1. Have ischemic ulcer.
2. Diagnosed with Buerger's disease.
3. Have a current or past history of life-threatening allergies.
4. Have been shown or are suspected to have cancer.
5. With concurrent proliferative intraocular neovascularization.
6. With poorly controlled diabetes mellitus.
7. With concurrent cardiac failure.
8. With untreated severe arrhythmia.
9. Have or are suspected to have interstitial pneumonia.
10. Have progressive hepatic disorders.
11. Have moderate or severe hepatic disorders. (1) aspartate aminotransferase or alanine aminotransferase >2.5 times the upper limit (2) Prothrombin time is 14 seconds or longer (3) Serum bilirubin >2.0 times the upper limit
12. Diagnosed with hepatic cirrhosis (classified as B or C on the Child-Pugh).
13. Have an inflammatory disease.
14. Treated with immunosuppressants or corticosteroids for the treatment of various inflammatory diseases or after organ transplantation.
15. Underwent extirpative surgery of a malignant tumor in the past 5 years.
16. Have had a cerebral hemorrhage or cerebral infarction in the past 6 months.
17. With blood diseases.
18. With moderate or severe renal dysfunction (CCr <40 mL/min)
19. With alcohol or drug dependence.
20. Pregnant/lactating female, or who wish or are suspected to be pregnant.
21. Positive HIV antibodies.
22. Took part in any other clinical studies or research in the past 30 days.
23. Have allergic to the antibiotics and/or the Ribavirin.
24. Not permitted to participate in this study by the principal investigator or sub-investigator for any other reasons.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-10 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Walking performance assessed by treadmill utilizing Gardner's method | 6 months
  Change rate from baseline in absolute claudication distance (%ACD) at 6 months Change of ACD from baseline at 6 months Change of peak walking time from baseline at 6 months Change of initial claudication distance (ICD) from baseline at 6 months Change of claudication onset time from baseline at 6 months

SECONDARY OUTCOMES:
NIRS measurement | Pre, day 14, 1, 2, 3, 4, 5, and 6 months
  Measurement of oxygen dynamics in the leg muscles by near infrared spectroscopy after a treadmill
Readministration | 6 months
  Proportion of subjects in whom readministration was not required
WIQ | Pre, 1, 3, and 6 months
  Evaluation of QOL based on the Walking Impairment Questionnaire (WIQ)
Clinical stage classifications | Pre, day 14, 1, 2, 3, 4, 5, and 6 months
  Time-course changes using clinical stage classifications (Fontaine classification, Rutherford classification)
ABI/TBI | Pre, day 14, 1, 3, and 6 months
  Ankle-brachial pressure index/ Toe-brachial pressure index
VAS | Pre, day 1, 2, 3, 5, 7, 14 and monthly until 6 months
  visual analogue scale (VAS) and pain at rest evaluated by the frequency of analgesic use
MACE | Monthly until 1 year after gene transfer
  Incidence of cardiovascular events (to be followed up to 5 years after administration)

CONTACTS AND LOCATIONS:
Overall Officials: Yoshikazu Yonemitsu, Study Chair — Kyushu University
Locations (4):
- Japan (4):
  - Matsuyama Red-Cross Hospital, Matsuyama, Ehime
  - Kyushu University Hospital, Fukuoka
  - Kyushu Central Hospital, Fukuoka
  - Morinomiya Hospital, Osaka

REFERENCES:
- [Background] Yonemitsu Y, Matsumoto T, Itoh H, Okazaki J, Uchiyama M, Yoshida K, Onimaru M, Onohara T, Inoguchi H, Kyuragi R, Shimokawa M, Ban H, Tanaka M, Inoue M, Shu T, Hasegawa M, Nakanishi Y, Maehara Y. DVC1-0101 to treat peripheral arterial disease: a Phase I/IIa open-label dose-escalation clinical trial. Mol Ther. 2013 Mar;21(3):707-14. doi: 10.1038/mt.2012.279. Epub 2013 Jan 15. PMID 23319060
- [Background] Matsumoto T, Tanaka M, Yoshiya K, Yoshiga R, Matsubara Y, Horiuchi-Yoshida K, Yonemitsu Y, Maehara Y. Improved quality of life in patients with no-option critical limb ischemia undergoing gene therapy with DVC1-0101. Sci Rep. 2016 Jul 15;6:30035. doi: 10.1038/srep30035. PMID 27418463